CLINICAL TRIAL: NCT05901103
Title: The Efficacy of Serratus Posterior Superior Intercostal Plane Block (SPSIPB) on Postoperative Pain and Total Analgesic Consumption in Patients Undergoing Video-assisted Thoracoscopic Surgery (VATS)
Brief Title: The Efficacy of SPSIPB on Postoperative Pain and Analgesic Consumption in Patients Undergoing VATS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cumhuriyet University (Other)
Responsible Party: Principal Investigator, Oguz Gundogdu, Assisstant Professor, Cumhuriyet University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: SPSIP block on VATS
Record Dates: First submitted 2023-06-01; First posted 2023-06-13 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Post Operative Pain
Keywords: serratus posterior superior intercostal plane block; video assisted thoracoscopic surgery; postoperative pain; regional anesthesia
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SPSIPB (Active Comparator): Serratus posterior superior intercostal plane block is the intervention used in this study. It was performed when the patient is in lateral decubitis position. A high frequency (7-12 MHz) linear transducer of the ultrasound device is placed at the spinae scapula level in the transverse plane, and the upper medial border of the scapula, the trapezius muscle, rhomboid muscle, serratus posterior superior muscle (SPSM) and the second and third ribs are visualized. The sonovisible needle is then advanced immediately medial to the scapula, aiming for the area between the second and third ribs in order to reach the fascial plane between the SPSM and intercostal muscles. After contact of the needle with the rib gently, 1-2mL of saline is used to confirm the correct plane, and a total of 30 mL of 0.25% bupivacaine is administered to the superficial to the intercostal muscle. PCA device was also performed to this group with the same protocol which was detailed in control arm.
  Interventions: Other: Serratus posterior superior intercostal plane block (SPSIPB)
- Control (No Intervention): Control group patients were not subjected to any block or local infiltration anesthesia (local anesthetic administration around the incision). Their postoperative pain was relieved with tramadol (intravenous analgesic drug) administration by using patient-controlled analgesia (PCA) device. Patient-controlled analgesia was achieved with tramadol hydrochloride at a concentration of 4 mg per 1 ml with the PCA device. The PCA device was configured to administer the patients boluses of 10 mg tramadol hydrochloride with a lockout time of 20 minutes, allowing a maximum of 4 pushes per hour. The total dose was standardized for all patients with a maximum daily dose of 400 mg and a maximum dose of 100 mg tramadol hydrochloride every 6 hours.

INTERVENTIONS:
Other: Serratus posterior superior intercostal plane block (SPSIPB) — Serratus posterior superior intercostal plane block is the intervention used in this study. It was performed when the patient is in lateral decubitis position. A high frequency (7-12 MHz) linear transducer of the ultrasound device is placed at the spinae scapula level in the transverse plane, and the upper medial border of the scapula, the trapezius muscle, rhomboid muscle, serratus posterior superior muscle (SPSM) and the second and third ribs are visualized. The sonovisible needle is then advanced immediately medial to the scapula, aiming for the area between the second and third ribs in order to reach the fascial plane between the SPSM and intercostal muscles. After contact of the needle with the rib gently, 1-2mL of saline is used to confirm the correct plane, and a total of 30 mL of 0.25% bupivacaine is administered to the superficial to the intercostal muscle.
  Arms: SPSIPB

SUMMARY:
The aim of this study is to investigate the postoperative analgesic efficacy of SPSIPB and its effect on opioid consumption in patients undergoing video-assisted thoracoscopic surgery (VATS).

DETAILED DESCRIPTION:
There were two randomized groups: Group S (SPSIPB) (n=12), Group C (no block) (n=12). All patients had standard general anesthesia. Group S had serratus posterior superior intercostal plane block (SPSIPB) with 0.25% bupivacaine (total volume of 30 ml) at the end of the surgery. Group Control had only tramadol for postoperative pain. Numerical rating scale (NRS) was used to assess postoperative pain on 1st, 6th, 12th and 24th hour after the surgery. Total tramadol consumption was calculated using patient-controlled analgesia (PCA) device.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients older than 18 years of age who underwent video-assisted thoracoscopic surgery (VATS) under general anesthesia and were American Society of Anesthesiologists (ASA) I-II-III according to the ASA risk classification.

Exclusion Criteria:

* Patients who did not give consent,
* patients with coagulopathy,
* patients with signs of infection at the block application site,
* patients using anticoagulants,
* patients with local anesthetic drug allergies,
* patients undergoing open surgery,
* patients with unstable hemodynamics,
* patients who could not cooperate during postoperative pain assessment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2023-03-29 (Actual); Primary Completion 2023-05-25 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Numerical rating scale (NRS) scores | Postoperative 24 hours
  Numerical rating scale is used for pain assessment. The scores of the numerical rating scale changes between 0 to 10 points. 10 points mean "the most severe pain that the patient ever had". 0 point means "there is no pain." Higher scores mean worse outcome.

SECONDARY OUTCOMES:
Total tramadol consumption | Postoperative 24 hours
  Postoperative analgesic (tramadol) need is measured by using patient-controlled analgesia (PCA) device.

CONTACTS AND LOCATIONS:
Locations (1):
- Sivas Cumhuriyet University, Sivas, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tulgar S, Ciftci B, Ahiskalioglu A, Bilal B, Sakul BU, Korkmaz AO, Bozkurt NN, De Cassai A, Torres AJ, Elsharkawy H, Alici HA. Serratus Posterior Superior Intercostal Plane Block: A Technical Report on the Description of a Novel Periparavertebral Block for Thoracic Pain. Cureus. 2023 Feb 3;15(2):e34582. doi: 10.7759/cureus.34582. eCollection 2023 Feb. PMID 36883093